CLINICAL TRIAL: NCT05574036
Title: Comparative Study Evaluating the Outcome of Febuxostat Versus Vitamin E in Hyperuricemia Patients With Non-alcoholic Steatohepatitis Without Cirrhosis
Brief Title: Comparative Study Between Febuxostat Versus Vitamin E in Non-alcoholic Steatohepatitis Patients With Hyperuricemia
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Hadier Mohammed El-Sheikh, Assistant lecturer of clinical pharmacy- Clinical pharmacy department- Faculty of pharmacy, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 34512/2/22
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2025-01-23 (Actual); Status verified 2025-01

CONDITIONS: Non Alcoholic Steatohepatitis; Hyperuricemia
Keywords: Hyperuricemic NAFLD; Elevated uric acid with fatty liver
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease; Hyperuricemia | interventions — Febuxostat; Tablets; Vitamin E

STUDY DESIGN:
Intervention Model Description: This study is randomized controlled, parallel and prospective 6-months duration study. Accepted patients will be randomized into 2 groups as the following:
  * Group 1 (Febuxostat group): 35 patients will receive 80 mg/day febuxostat for 6 months.
  * Group 2 (Control group): 35 patients will receive Vitamin E 400 mg twice daily for 6 months.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group 1 Febuxostat group (Active Comparator): 35 non alcoholic steatohepatitis hyperuricemic patients receiving Febuxostat 80 mg once daily for 6 months duration
  Interventions: Drug: Febuxostat 80 MG Oral Tablet
- Group 2 vitamin E group (Active Comparator): 35 non alcoholic steatohepatitis Hyperuricemic patients receiving vitamin E 400 mg twice daily for 6 months duration
  Interventions: Drug: vit E

INTERVENTIONS:
Drug: Febuxostat 80 MG Oral Tablet — Febuxostat used as 80 mg oral tablet once daily for 6 months
  Other Names: Andouristat 80 mg, Staturic 80 mg
  Arms: Group 1 Febuxostat group
Drug: vit E — Vitamin E used as 400 mg soft gelatin capsules twice daily for 6 months
  Other Names: Vitamin E 400 mg
  Arms: Group 2 vitamin E group

SUMMARY:
This study aims at evaluating and comparing the protective outcomes of using Febuxostat versus Vitamin E in Hyperuricemia non-alcoholic steatohepatitis patients without cirrhosis. The intervention is 6-months duration and the study will assess the efficacy of either drug as fibrosis improvement (≥ 1 stage) with no worsening of NASH or NASH resolution with no worsening of fibrosis with the study considered successful if either 1ry end point is met. Also, assessment of biochemical markers related to steatosis, inflammation, oxidative stress, insulin resistance and liver fibrosis will be done.

DETAILED DESCRIPTION:
Nonalcoholic fatty liver disease (NAFLD) is defined as the accumulation of excessive fat in the liver in the setting of no significant alcohol consumption and the absence of any secondary cause. NAFLD has reached epidemic proportions and currently affects 20-40% of the general population. In recent years, along with the increasing trend of obesity and type 2 diabetes, NAFLD has become one of the most common chronic liver diseases worldwide. The spectrum of the disease ranges from simple steatosis to hepatocellular injury with inflammatory infiltration characterized as nonalcoholic steatohepatitis (NASH) that may eventually progress to liver fibrosis, cirrhosis and hepatocellular carcinoma. Despite significant disease burden and mortality associated mainly with advanced disease, i.e., NASH and fibrosis, there is currently no approved medication for NASH, therefore, lifestyle modifications remain the mainstay of treatment. What is the pathogenesis of NAFLD? Although the proposal of "two hits" involving insulin resistance (IR) and oxidative stress has been well accepted, the mechanism of NAFLD was thought very complex and still remained unclearly.

Besides metabolic syndrome-related conditions, hyperuricemia has also been linked to NASH. Several epidemiological studies have demonstrated that patients with NASH have significantly higher serum uric acid (UA) levels relative to controls, and elevated serum UA levels are an independent risk factor for NAFLD. Notably, UA itself has been reported to promote de novo lipogenesis and induce IR, both in vivo and in vitro, through increased NADPH oxidase (NOX)-mediated reactive oxygen species (ROS) generation and activation of the Nucleotide-binding and oligomerization domain (NOD-like) receptor family pyrin domain containing 3 (NLRP3) inflammasome. It is thought that hyperuricemia in NAFLD is primarily due to increased expression and/or activity of hepatic xanthine oxidase (XO). These observations indicate that hyperuricemia plays a causative role in the development of NASH.

The xanthine oxidase (XO) inhibitor, febuxostat, decreases free fatty acids-induced fat accumulation in the liver of high-fat diet containing trans-fatty acids (HFDT) fed mice. It was further found that the underlying mechanism is related to the reduction in expression of NLRP3 and improved insulin resistance. This finding highlights the possible molecular pathways involving NLRP3 activation for management of ROS and IR. In conclusion, febuxostat may be a promising potential treatment for patients with NASH.

It is acknowledged that vitamin E is the major lipid-soluble chain-breaking antioxidant found in the human body. In addition to its anti-oxidative properties, molecules of vitamin E family exert anti-atherogenic and anti-inflammatory activities. According to American Association for the Study of Liver Diseases (AASLD) and National Institute for Health and Care Excellence (NICE) guidelines, vitamin E is approved at a dose of 800 IU/day in adults with biopsy-proven NASH.

Therefore, This study aims at evaluating and comparing the protective outcomes of using Febuxostat versus Vitamin E in hyperuricemic NASH patients without cirrhosis.

The primary endpoint of this 6-months study would be fibrosis improvement (≥

1 stage) with no worsening of NASH or NASH resolution with no worsening of fibrosis with the study considered successful if either 1ry end point is met.

The secondary endpoint of this study is improvement of biochemical markers related to steatosis, inflammation, oxidative stress, insulin resistance and liver fibrosis.

Study Population:

* This study is conducted on 60 patients diagnosed with Hyperuricemic NASH according to the study protocol.
* Patients has been recruited from Tropical Medicine and Infectious Diseases Department, Tanta University Hospital, Tanta, Egypt.
* The study was approved by the Research Ethics Committee of Tanta University.
* All patients have provided signed written informed consent and agreed to comply with the study protocol.
* All data of the patients will be private and confidential.
* Any unexpected risks appeared during the course of the research was cleared to the patients and the ethical committee on time.

This study is randomized controlled, parallel and prospective 6-months duration study. Accepted patients was randomized into 2 groups as the following:

* Group 1 (Febuxostat group): 30 patients will receive 80 mg/day febuxostat for 6 months.
* Group 2 (Control group): 30 patients will receive Vitamin E 400 mg twice daily for 6 months.

Any side effects will be reported and graded according to common terminology criteria for adverse events version 5.00 (CTCAE). Any potential drug interactions between administered drugs is monitored for each patient and corrective actions is taken.

Statistical Analysis

* All data will be represented as mean ± slandered deviation (SD).
* Unpaired Student's t-test will be used to compare data between the two groups.
* Paired Student's t-test will be used to compare data within the same group before and after treatment with the studied medications.
* Chi-square test will be used for statistical analysis of nominal data.
* The statistical analysis will be carried out using Statistical Package for the Social Sciences (SPSS) statistical package version 27.0 (December 2020), IBM (International Business Machines) corporation software group, USA.
* The level of significance will be set at P< 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged ≥18 years.
* All patients are diagnosed to have fatty liver grading 1, 2 or 3 on abdominal ultrasound with Hepatic steatosis index > 36 to be considered as a NAFLD patient.
* Serum uric acid level ≥ 6 mg/dl.
* Confirmed diagnosis of NASH using at least three of the following non-invasive tests:
* HAIR score
* Fibroscan detecting steatosis with F0-3 fibrosis stage
* Cytokeratin-18 >240 U/L
* Mild to moderate elevation of serum aminotransferases (>2 but <5 times upper normal limit)

Exclusion Criteria:

* Current or history of significant alcohol consumption.
* Use of drugs historically associated with nonalcoholic fatty liver disease (NAFLD) (amiodarone, methotrexate, systemic glucocorticoids, tetracyclines, tamoxifen, estrogens at doses greater than those used for hormone replacement, anabolic steroids, valproic acid, and other known hepatotoxins).
* Prior or planned bariatric surgery.
* Patients with Hemoglobin A1c 9.5% or higher.
* Evidence of other forms of chronic liver disease as Hepatitis B, Hepatitis C, Wilson's disease, Alpha-1-antitrypsin(A1AT) deficiency, Hemochromatosis, drug-induced liver disease.
* Serum creatinine of 2.0 mg/dL or greater.
* Pregnancy, planned pregnancy, potential for pregnancy and unwillingness to use effective birth control during the trial and breast feeding.
* Use of other drugs known to have possible positive effects on steatosis.
* Patients on oral anticoagulants as warfarin.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in fibrosis stage; fibrosis improvement (≥ 1 stage), with no worsening of NASH, detected by fibroscan device | 6 months
  Patients will undergo fibroscan testing prior to the initiation of the intervention and after 6 months of receiving the drug therapy to detect fibrosis improvement
Change from baseline NASH condition at 6 months; NASH resolution, with no worsening of fibrosis, with the study considered successful if either 1ry end point is met. | 6 months
  Patients will undergo assessment of serum aminotransferases prior to the initiation of the intervention and after 6 months of receiving the drug therapy to detect NASH resolution
Change from baseline steatosis stage at 6 months detected by Fibroscan device | 6 months
  Patients will undergo fibroscan testing prior to the initiation of the intervention and after 6 months of receiving the drug therapy to detect steatosis improvement

SECONDARY OUTCOMES:
Change in serum level of Nucleotide-binding and oligomerization domain (NOD-like) receptor family pyrin domain containing 3 inflammasome(NLRP3) | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate NODlike receptor family pyrin domain containing 3 inflammasome(NLRP3)
Change in serum level of Malondialdehyde (MDA) | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate Malondialdehyde (MDA)
Change in serum uric acid | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate serum uric acid
Change in fasting insulin with calculation of Homeostasis Model Assessment (HOMA-IR). | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate fasting insulin with calculation of Homeostasis Model Assessment (HOMA-IR).
Change in serum level of cytokeratin-18 (CK-18) | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate cytokeratin-18 (CK-18)
Change in serum level of Total lipid profile (Total cholesterol, High density lipoprotein cholesterol and Triglycerides) with calculation of Low density lipoprotein. | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate Total cholesterol, High density lipoprotein cholesterol and Triglycerides with calculation of Low density lipoprotein.
Change in serum level of Liver enzymes; Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alk.Phosphatase (ALP) and Gamma-glutamyl transferase (GGT) | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate Alanine aminotransferase (ALT), Aspartate aminotransferase (AST), Alk. Phosphatase (ALP) and Gamma-glutamyl transferase (GGT)
Change in serum level of tissue inhibitor of metalloproteinase-1 (TIM-1) | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate tissue inhibitor of metalloproteinase-1(TIM-1)
Change in serum urea and creatinine. | 6 months
  Blood samples will be collected at baseline and after 6 months of receiving the intervention therapy to evaluate Serum urea and creatinine.

CONTACTS AND LOCATIONS:
Overall Officials: Hadier m. El-sheikh, Principal Investigator — Department of Clinical pharmacy, Faculty of Pharmacy, Tanta university
Locations (1):
- Department of Tropical Medicine and Infectious Diseases, Faculty of Medicine,Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available

REFERENCES:
- [Background] El Hadi H, Vettor R, Rossato M. Vitamin E as a Treatment for Nonalcoholic Fatty Liver Disease: Reality or Myth? Antioxidants (Basel). 2018 Jan 16;7(1):12. doi: 10.3390/antiox7010012. PMID 29337849
- [Background] Afzali A, Weiss NS, Boyko EJ, Ioannou GN. Association between serum uric acid level and chronic liver disease in the United States. Hepatology. 2010 Aug;52(2):578-89. doi: 10.1002/hep.23717. PMID 20683957
- [Background] Zhu Y, Hu Y, Huang T, Zhang Y, Li Z, Luo C, Luo Y, Yuan H, Hisatome I, Yamamoto T, Cheng J. High uric acid directly inhibits insulin signalling and induces insulin resistance. Biochem Biophys Res Commun. 2014 May 16;447(4):707-14. doi: 10.1016/j.bbrc.2014.04.080. Epub 2014 Apr 21. PMID 24769205
- [Background] Tang W, Mu J, Chen QI, Li X, Liu H. The involvement and mechanism of febuxostat in non-alcoholic fatty liver disease cells. J Biol Regul Homeost Agents. 2018 May-Jun;32(3):545-551. PMID 29921379
- [Background] Chalasani N, Younossi Z, Lavine JE, Charlton M, Cusi K, Rinella M, Harrison SA, Brunt EM, Sanyal AJ. The diagnosis and management of nonalcoholic fatty liver disease: Practice guidance from the American Association for the Study of Liver Diseases. Hepatology. 2018 Jan;67(1):328-357. doi: 10.1002/hep.29367. Epub 2017 Sep 29. No abstract available. PMID 28714183
- [Derived] El-Sheikh H, El-Haggar S, Badawi R, Habba E. Comparative efficacy of febuxostat and vitamin E in the management of MASLD: Insights from a randomized parallel clinical study. Eur J Pharmacol. 2025 Aug 5;1000:177735. doi: 10.1016/j.ejphar.2025.177735. Epub 2025 May 16. PMID 40383220
- See also: Effects of Febuxostat for Lowering Uric Acid in NAFLD Patients With Gout — https://www.clinicaltrials.gov/ct2/show/NCT04772352
- See also: Vitamin E and NAFLD — https://www.mayoclinic.org/drugs-supplements-vitamin-e/art-20364144